CLINICAL TRIAL: NCT00272714
Title: A Phase II, Randomized, Double-Blind, Two-Dose, Placebo-Controlled Multicentre Study of 4-Hydroxy Tamoxifen Gel for Cyclical Mastalgia in Otherwise Healthy Pre-Menopausal Women With Regular Menstrual Cycles.
Brief Title: Study of Afimoxifene Gel to Treat Cyclic Mastalgia in Premenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASCEND Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01-4OHT-02
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2013-07

CONDITIONS: Cyclic Breast Pain, Cyclic Mastalgia
Keywords: breast pain, tenderness, benign breast conditions
MeSH Terms: conditions — Mastodynia | interventions — afimoxifene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Afimoxifene (0.057%) in hydroalcoholic gel

SUMMARY:
The purpose of this study is to evaluate the efficacy of two doses of 4-hydroxy tamoxifen (4-OHT) compared with placebo on the intensity of cyclic mastalgia in pre-menopausal women with regular menstrual cycles who are not taking oral contraceptives.

DETAILED DESCRIPTION:
This study is a Phase II, randomised, double-blind, placebo-controlled, two-dose, multicentre trial of 4-OHT gel in approximately 130 otherwise healthy pre-menopausal women with a history of cyclical mastalgia, peaking during the second half of the menstrual cycle and decreasing significantly with the onset of menstruation, during the four months prior to study entry.

The primary efficacy endpoint in this study is change in change in average pain Visual Analog Scale (VAS) scores for the seven worst pain scores within a cycle, from baseline to the fourth cycle after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* A woman is eligible for this study if she:

  * is pre-menopausal and at least 18 years of age.
  * has a history of cyclical mastalgia for each of the four months prior to study entry.
  * moderate or severe mastalgia as determined by >40 mm on the VAS for ≥7 days per cycle in the second part of the cycle, i.e. 13 days prior to menses and the first two days of the next cycle with a substantial decrease during the two weeks following the onset of menses, assessed during the two month run-in period.
  * has a history of regular menstrual cycles of 28 plus/minus 3 days.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2003-03; Primary Completion 2004-03 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) scores for the seven worst scores within a cycle, from baseline to the forth cycle after treatment

SECONDARY OUTCOMES:
Change from baseline in average VAS pain scores for the seven worst pain scores within a cycle over all cycles
Change from baseline in average VAS pain scores over all scores over all cycles
Change from baseline in the number of nominal days of breast pain (NDBP) over all cycles using the Cardiff Breast Pain Chart.
Physician's global assessment of pain.
Physician's clinical evaluation of mastalgia (tenderness determined by palpation).
Physician's clinical evaluation of mastalgia (nodularity).
Patient's global assessment of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Mansel, MD, Principal Investigator — University of Wales College of Medicine